CLINICAL TRIAL: NCT05272696
Title: Induction Therapy With Nab-paclitaxel, Cisplatin and Pembrolizumab in Untreated Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Pembrolizumab and Induction Chemotherapy in Locally Advanced HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, MA HAIQING, chief physician, Guangdong Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INDUCTION THERAPY
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — 130-nm albumin-bound paclitaxel; Cisplatin; Surgical Procedures, Operative; Chemoradiotherapy, Adjuvant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): All enrolled patients will receive two cycles of chemotherapy consisting of nab-paclitaxel (260 mg/m² on days 1), cisplatin (75 mg/m² on days 1), and Pembrolizumab (200 mg on days 1). Each cycle is repeated every 21 days.
  After induction therapy, patients with PR but the maximum diameter of tumor > 3cm or SD or PD can receive surgery directly. After surgery, adjuvant CRT will be given for patients with high-risk factors.
  After induction therapy, patients with PR and maximum tumor diameter ≤ 3cm or CR evaluated by MDT after 2 courses induction therapy can receive CRT. Evaluation was performed 3 months after CRT. After MDT discussion, patients with high-risk factors need maintenance treatment.
  Interventions: Drug: Nab-paclitaxel, cisplatin and Pembrolizumab combination; Procedure: surgery; Radiation: Adjuvant Chemoradiotherapy; Drug: Radical concurrent chemoradiotherapy

INTERVENTIONS:
Drug: Nab-paclitaxel, cisplatin and Pembrolizumab combination — Pembrolizumab in combination with Nab-paclitaxel and cisplatin as induction therapy
Procedure: surgery — Patients with PR but the maximum diameter of tumor > 3cm or SD or PD can receive surgery directly.
Radiation: Adjuvant Chemoradiotherapy — After surgery, adjuvant Chemoradiotherapy or radiotherapy will be given for patients with high-risk factors.
Drug: Radical concurrent chemoradiotherapy — Patients with PR and maximum tumor diameter ≤ 3cm or CR evaluated by MDT after 2 courses induction therapy can receive Radical concurrent chemoradiotherapy. Evaluation was performed 3 months after CRT. After MDT discussion, patients with high-risk factors need maintenance treatment.

SUMMARY:
To study induction therapy with Nab-paclitaxel, Cisplatin and Pembrolizumab in patients with Locally Advanced HNSCC.

DETAILED DESCRIPTION:
This study is a non-randomized, single-arm, single-institutional phase II study including patients with Locally Advanced Head and Neck Squamous Cell Carcinoma eligible for resection. Nab-paclitaxel (260 mg/m² IV), cisplatin (75 mg/m² IV), and Pembrolizumab (200 mg IV) will be administered for two cycles of three weeks duration each. Surgery or CRT will be performed after induction therapy. Patients with PR and maximum tumor diameter ≤ 3cm or CR evaluated by MDT after 2 courses induction therapy can receive CRT. Evaluation was performed 3 months after CRT. After MDT discussion, patients with high-risk factors need maintenance treatment. Patients with PR but the maximum diameter of tumor > 3cm or SD or PD can receive surgery directly. After surgery, adjuvant CRT will be given for patients with high-risk factors. Objective response rate, safety, and rate of organ preservation will be the primary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed Head and Neck Squamous Cell Carcinoma (oral cavity, oropharynx, laryngeal and hypopharynx) with locoregionally-advanced disease stage III or IVA without metastasis , previously untreated (AJCC 8th) and had at least one tumour lesion measurable per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
2. Measurable disease based on RECIST 1.1
3. ECOG performance status 0-1
4. Men and women, Age ≥18 and ≤ 70 years at the time of signing informed consent,
5. Adequate hepatic, cardiac and renal function as demonstrated by 1) Hematology: ANC≥1.5×10^9 /L, HGB≥9 g/dL, PLT≥80×10^9 /L; 2) Renal: Serum creatinine < 1.5x ULN or CrCl > 60mL/min; 3) Hepatic: Total Bilirubin ≤ 1.5 x ULN, AST/ALT ≤ 2.5 x ULN and ALP≤5 x ULN.
6. Female subjects of childbearing potential should have a negative pregnancy test result within 28 days prior to enrollment. If the result is more than 7 days before receiving the first dose of study medication, a urine pregnancy test is required for verification.
7. Voluntary informed consent, joining the study with good compliance

Exclusion Criteria:

1. Active, known, or suspected autoimmune disease or Type I diabetes or hypothyroidism requiring hormone replacement therapy and skin diseases requiring systemic treatment.
2. currently received systemic steroid therapy with dose superior to 10 mg/day of prednisone or equivalent or any other form of immunosuppressive therapy within 14 days prior to the enrollment
3. Has known active Hepatitis B (e.g., HBsAg reactive and HBV DNA≥1×10^4 copies /mL) or Hepatitis C or HIV
4. Active pulmonary tuberculosis (TB) infection was judged according to chest X-ray examination/CT, sputum examination and clinical physical examination.
5. Patients with severe heart disease include congestive heart failure, uncontrollable high-risk arrhythmias, unstable angina pectoris, myocardial infarction, and intractable hypertension.
6. Pregnant or breastfeeding women.
7. The patient (male or female) has the possibility of fertility, but is unwilling or does not take effective contraceptive measures.
8. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device
9. Has had another known invasive malignancy or unresectable cancer.
10. Received a live vaccine within 30 days of planned start of study therapy.
11. History or current evidence of any condition, therapy, or laboratory abnormality that might influence the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 24 months
  Objective response rate (ORR) will be determinated by evaluation of Complete Response (CR) and Partial Response (PR)
Evaluation of Safety | 24 months
  Toxicity will be evaluated according to NCI-CTCAE v4.03
Rate of organ preservation | 24 months
  After two courses of induction treatment, MDT discussed whether to accept surgical treatment or concurrent chemoradiotherapy, and the proportion of patients whose organ function can be preserved after treatment.

SECONDARY OUTCOMES:
overall survival (OS) | 24 months
  Defined from date of registration to date of first documentation of death from any cause or censored at the date of the last follow-up.
progression-free survival (PFS) | 24 months
  Defined from date of registration to date of first documentation of progression or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No